CLINICAL TRIAL: NCT06039384
Title: A Phase 1 Study of INCB099280 in Combination With Adagrasib in Adults With Advanced Solid Tumors Harboring a KRASG12C Mutation
Brief Title: A Study of INCB099280 in Combination With Adagrasib in Adults With Advanced Solid Tumors Harboring a KRASG12C Mutation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This was a strategic business decision. There were no safety concerns contributing to this decision.
Sponsor: Incyte Corporation (Industry)
Collaborators: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCB99280-204; 2023-503223-26-00 (Registry Identifier: EU CT number)
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumors
Keywords: KRASG12C mutation; non-small cell lung cancer (NSCLC); colorectal cancer (CRC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms | interventions — adagrasib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Finding (Experimental): INCB099280 administered in combination with adagrasib in participants with previously treated KRAS glutamine to cysteine mutation at codon 12 (KRASG12C) mutant advanced solid tumors, will be evaluated to identify dose(s) for further evaluation in the dose expansion phase of the study.
  Interventions: Drug: INCB099280; Drug: adagrasib
- Part 2: Dose Expansion (Experimental): Up to 80 participants will be enrolled in 1 of 2 disease-specific cohorts: Cohort A: previously treated KRASG12C mutated non-small cell lung cancer (NSCLC) Cohort B: previously treated KRASG12C-mutated colorectal cancer (CRC). Up to 3 doses may be selected from Part 1: Dose Finding for the Part 2: Dose Expansion.
  Interventions: Drug: INCB099280; Drug: adagrasib

INTERVENTIONS:
Drug: INCB099280 — Administered as specified in the treatment arm description
Drug: adagrasib — Administered as specified in the treatment arm description
  Other Names: KRAZATI

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of INCB099280 in combination with adagrasib and to establish the MTD or identify RDE(s) for the combination of INCB099280 and adagrasib.

ELIGIBILITY:
Inclusion Criteria:

* KRASG12C-mutated solid malignancy determined by a sponsor-approved assay using either tumor tissue or ctDNA.
* Histologically confirmed malignant solid tumor with locally advanced and/or metastatic disease.

  * Only participants with NSCLC will be enrolled into Part 2 Cohort A.
  * Only participants with CRC will be enrolled into Part 2 Cohort B.
* Part 1: Disease progression on or after at least 1 prior systemic treatment.
* Part 2 (Cohort A - NSCLC): Received an anti-PD-(L)1-containing regimen and platinum based chemotherapy regimen either concurrently or sequentially
* Part 2 (Cohort B - CRC): Received at least 1 line of systemic therapy that includes the combination of fluoropyrimidine-based chemotherapy (in combination with oxaliplatin and/or irinotecan) and either a vascular endothelial growth factor-targeting monoclonal antibody or an anti-epidermal growth factor receptor monoclonal antibody (if RAS wild type). Participants with MSI-H/dMMR CRC must also have received a prior immune checkpoint inhibitor approved for this indication.
* Measurable disease according to RECIST v1.1.
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* Estimated life expectancy > 3 months.
* Willingness to avoid pregnancy.

Exclusion Criteria:

* Known additional malignancy that is progressing or requires active treatment.
* Central nervous system (CNS) metastases requiring treatment and/or leptomeningeal disease.
* Part 2 only: Prior treatment with an approved or investigational agent targeting KRASG12C.
* Toxicity from prior therapy that has not recovered to protocol-defined limits.
* Received thoracic radiation of > 30 Gy within 6 months of the first dose of study treatment.
* Participation in another interventional clinical study.
* History or evidence of interstitial lung disease, including noninfectious pneumonitis.
* Presence of gastrointestinal condition that may affect drug absorption.
* Active autoimmune disease requiring systemic treatment, including corticosteroids exceeding a daily dose of 10 mg of prednisone or equivalent.
* Diagnosis of immunodeficiency or receiving chronic systemic steroid therapy exceeding a daily dose of 10 mg of prednisone or equivalent.
* Active infection requiring systemic therapy.
* History of organ transplantation, including allogeneic stem cell transplantation.
* Receipt of systemic antibiotics within 28 days of the first dose of study treatment.
* Probiotic usage is prohibited during screening and throughout the study treatment period.
* Received a live vaccine within 28 days of the planned start of study drug.
* Laboratory values outside the Protocol-defined ranges.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-12-28 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of participants with Dose Limiting Toxicities (DLTs) | Up to 28 days
  Dose-limiting toxicity will be defined as the occurrence of any of the toxicities as per protocol.
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to 2 years and 90 days
  Defined as adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug.
Number of participants with TEAEs leading to dose modification or discontinuation | Up to 2 years and 90 days
  Number of participants with TEAEs leading to dose modification or discontinuation.

SECONDARY OUTCOMES:
INCB099280 and adagrasib plasma concentrations. | Up to 2 years
  PK parameters will be calculated from the blood plasma concentrations of INCB099280 and adagrasib using standard noncompartmental (model independent) PK methods.
Objective response rate (ORR) | Up to 2 years
  Defined as having a best overall response of complete response (CR) or partial response (PR) assessed per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by the investigator.
Disease Control Rate (DCR) | Up to 2 years
  Defined as having a best overall response of CR, PR, or stable disease (SD) ≥ 15 weeks (from the start of treatment) assessed per RECIST v1.1 by the investigator.
Duration of Response (DOR) | Up to 2 years
  Defined as the time from the first CR or PR until disease progression (assessed per RECIST v1.1 by the investigator) or death from any cause, whichever occurs earlier.
Progression-free survival (PFS) | Up to 12 months
  Defined as absence of disease progression (assessed per RECIST v1.1 by the investigator) or death from any cause from start of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (14):
- United States (5):
  - Valkyrie Clinical Trials, Los Angeles, California
  - Banner Md Anderson Cancer Center, Greeley, Colorado
  - Henry Ford Health System, Detroit, Michigan
  - Mary Crowley Cancer Research Centers McCrc Headquarters, Dallas, Texas
  - Inova Schar Cancer Institute, Falls Church, Virginia
- Italy (3):
  - Fondazione Del Piemonte Per L Oncologia Ircc Candiolo, Candiolo
  - Irccs Istituto Clinico Humanitas, Rozzano
  - Centro Ricerche Cliniche Di Verona (Crc), Verona
- Spain (4):
  - Hospital Hm Nou Delfos, Barcelona
  - Hospital General Universitario Vall D Hebron, Barcelona
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón
  - Hospital Universitario Virgen Macarena, Seville
- United Kingdom (2):
  - Guys Hospital, London
  - Hammersmith Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency